CLINICAL TRIAL: NCT04057014
Title: A Prospective Study of Immediate Versus Delayed Treatment of Odontogenic Infections
Brief Title: Immediate Versus Delayed Treatment of Odontogenic Infections
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding available for the activity
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Keri Discepolo, Associate Dentist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00030880
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Focal Infection, Dental
Keywords: Dentistry; Antibiotic; Penicillin; pediatrics
MeSH Terms: conditions — Focal Infection, Dental | interventions — Amoxicillin; Tooth Extraction

STUDY DESIGN:
Intervention Model Description: Prospective partially randomized parallel study groups clinical trial investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Extraction Only (Active Comparator): Immediate extraction of infected tooth without antibiotic prescription.
  Interventions: Procedure: Tooth extraction
- Average Dose Antibiotic (Experimental): Average dose antibiotic therapy(25 mg/kg/day in divided doses every 12 hours (maximum 875 mg/dose)) for 10 days and receive tooth extraction on day 10 (25 patients). (*given the average weight of a 12 year old is 45 kilos, we do not expect that we will reach the maximum dose in this group)
  Interventions: Drug: Amoxicillin; Procedure: Tooth extraction
- High Dose Antibiotic (Experimental): High dose antibiotic therapy (45 mg/kg/day in divided doses every 12 hours (maximum 875 mg/dose)) for 5 days and receive tooth extraction on day 10 (25 patients)
  Interventions: Drug: Amoxicillin; Procedure: Tooth extraction

INTERVENTIONS:
Drug: Amoxicillin — Antibiotic given at different dosages and durations.
  Other Names: Amoxil
  Arms: Average Dose Antibiotic; High Dose Antibiotic
Procedure: Tooth extraction — Removal of infected tooth on first day of study, this approach does not require an antibiotic drug.
  Other Names: Exodontia

SUMMARY:
The objective of this study is to compare the physiologic resolution of dental infections between immediate tooth extraction (control group) and administration of systemic antibiotics and delayed extraction (study groups 1 and 2). A secondary objective is two compare two different antibiotic regimens in the delayed extraction groups (study group 1 and 2).

DETAILED DESCRIPTION:
This is a prospective partially randomized clinical trial. Patients 2-11 years old who have a vestibular swelling associated with an odontogenic infection are being studied. Subjects will self-select into the control or study group. All subjects will be offered to have the tooth extracted on the day of diagnosis, and if this treatment is chosen they will join the control group (group 1). Subjects who defer treatment will be placed on amoxicillin and will be placed into the study group. The study group will be randomized into two parallel study groups that either have average dose antibiotics for 10 days (group 2), or maximum dose antibiotics for 5 days (group 3).

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the dental clinic or Boston Children's Hospital emergency room
* Odontogenic origin associated with a primary tooth and limited to the buccal vestibule only
* Ages of 2-11 years old
* Primary Caregiver present
* English speaking
* American Society of Anesthesiologists (ASA) classification of I
* None or current systemic antibiotic therapy regimen < 24 hours
* Able to take medication orally
* Those patients who choose to participate in the study

Exclusion Criteria:

* Infection that has spread beyond the buccal vestibule, or not detectable
* Infection is associated with a permanent adult tooth
* Ages of <2 years old or >11 years old
* American Society of Anesthesiologists classification of II or greater or poor general health.
* Renal impairment
* Immunosuppressive disease
* Recent antibiotic therapy in the last 1 to 30 days
* Allergy to penicillin
* Unable to take oral medications
* Decline participation

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Change in diagnosis | Infection will be monitored at days 0, 5, 10 and 20.
  Tooth infection not clinically detectable

SECONDARY OUTCOMES:
Measure of pediatric oral health-related quality of life: the POQL | Survey of quality of life at days 0, 5, 10 and 20.
  Quality of life compared between arms. Pediatric Oral Health Quality of Life (PQOL) clustered into four dimensions - Physical Functioning, Role Functioning, Social Functioning and Emotional Functioning. It was designed to be used in high risk, low resource, populations with greater health disparities. Specifically we are looking significant difference between the study groups that is at least 2 standard errors from the control group. If there are not two deviations to discriminate between scales would indicate a non-significant finding.

CONTACTS AND LOCATIONS:
Overall Officials: Keri Discepolo, DDS, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participant data.

REFERENCES:
- [Background] Dodson TB, Perrott DH, Kaban LB. Pediatric maxillofacial infections: a retrospective study of 113 patients. J Oral Maxillofac Surg. 1989 Apr;47(4):327-30. doi: 10.1016/0278-2391(89)90331-5. PMID 2926541
- [Background] Biederman GR, Dodson TB. Epidemiologic review of facial infections in hospitalized pediatric patients. J Oral Maxillofac Surg. 1994 Oct;52(10):1042-5. doi: 10.1016/0278-2391(94)90172-4. PMID 8089789
- [Background] Rush DE, Abdel-Haq N, Zhu JF, Aamar B, Malian M. Clindamycin versus Unasyn in the treatment of facial cellulitis of odontogenic origin in children. Clin Pediatr (Phila). 2007 Mar;46(2):154-9. doi: 10.1177/0009922806289431. PMID 17325089
- [Background] Warnke PH, Becker ST, Springer IN, Haerle F, Ullmann U, Russo PA, Wiltfang J, Fickenscher H, Schubert S. Penicillin compared with other advanced broad spectrum antibiotics regarding antibacterial activity against oral pathogens isolated from odontogenic abscesses. J Craniomaxillofac Surg. 2008 Dec;36(8):462-7. doi: 10.1016/j.jcms.2008.07.001. Epub 2008 Aug 29. PMID 18760616
- [Background] Kara A, Ozsurekci Y, Tekcicek M, Karadag Oncel E, Cengiz AB, Karahan S, Ceyhan M, Celik MO, Ozkaya-Parlakay A. Length of hospital stay and management of facial cellulitis of odontogenic origin in children. Pediatr Dent. 2014 Jan-Feb;36(1):18E-22E. PMID 24717702
- [Background] Lin YT, Lu PW. Retrospective study of pediatric facial cellulitis of odontogenic origin. Pediatr Infect Dis J. 2006 Apr;25(4):339-42. doi: 10.1097/01.inf.0000216202.59529.3d. PMID 16567986
- [Background] Huntington NL, Spetter D, Jones JA, Rich SE, Garcia RI, Spiro A 3rd. Development and validation of a measure of pediatric oral health-related quality of life: the POQL. J Public Health Dent. 2011 Summer;71(3):185-93. PMID 21972458
- [Background] Thikkurissy S, Rawlins JT, Kumar A, Evans E, Casamassimo PS. Rapid treatment reduces hospitalization for pediatric patients with odontogenic-based cellulitis. Am J Emerg Med. 2010 Jul;28(6):668-72. doi: 10.1016/j.ajem.2009.02.028. Epub 2010 Apr 2. PMID 20637381